CLINICAL TRIAL: NCT02128243
Title: Randomized Controlled Trial of S-1 Maintenance Therapy in Metastatic Esophagogastric Cancer
Brief Title: Trial of S-1 Maintenance Therapy in Metastatic Esophagogastric Cancer
Acronym: MATEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry); Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-YMO-0111; 2013-002742-37 (EudraCT Number)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Unresectable, Locally Advanced or Metastatic, Adenocarcinoma of the Stomach, or of the Gastro Esophageal Junction; Gastric Neoplasm; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma; Gastric Adenocarcinoma; Esophageal Neoplasms
MeSH Terms: conditions — Neoplasm Metastasis; Stomach Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — tegafur-gimeracil-oteracil; Oxaliplatin; Leucovorin; Fluorouracil; Cisplatin; S 1 (combination); Epirubicin; Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: De-escalation therapy (Experimental): Patients in Arm A will continue with S-1 de-escalation phase starting at week 13 until disease progression, toxicities requiring discontinuation, withdrawal of consent, pregnancy, death or lost to follow up whichever occurs first. In patients with drug-related severe toxicity S-1 dose will be adjusted or study treatment will be terminated.
  Interventions: Drug: S-1 de-escalation
- Arm B: Chemotherapy by Investigator's choice (Experimental): Patients in Arm B will continue to receive the same polychemotherapy as during induction therapy until tumor progression, toxicities requiring discontinuation, withdrawal of consent, pregnancy, death or loss to follow up whichever occurs first.
  Interventions: Drug: Chemotherapy by Investigator's choice

INTERVENTIONS:
Drug: S-1 de-escalation — S-1 30 mg/m² bid d1-14 q21d
  Other Names: Teysuno
  Arms: Arm A: De-escalation therapy
Drug: Chemotherapy by Investigator's choice — Polychemotherapy administration as in induction therapy consists of a platinum and fluoropyrimidine compound as well as optional a taxane / an anthracycline compound.
  Two-Drug combinations:
  FLO / mod. FOLFOX-6; Cisplatin, S-1; Cisplatin, 5-FU; Cisplatin, Capecitabine (XP)
  Three-drug combinations:
  EOX/EOF FLOT
  Other Names: FLO regimen; - Oxaliplatin 85 mg/m²; - Leucovorin 200 mg/m²; - 5-Fluorouracil 2600 mg/m²; mod. FOLFOX-6 regimen; - Leucovorin 400 mg/m²; - 5-Fluorouracil 400 mg/m²; - 5-Fluorouracil 2400 mg/m²; Cisplatin / S-1; - Cisplatin 75 mg/m²; - S-1 25mg/m²; EOX/EOF; - Epirubicin 50 mg/m²; - Oxaliplatin 130 mg/m²; - Capecitabine 625 mg/m²; FLOT; - Docetaxel 50 mg/m²; - Leucovorin 200 mg/mg²; Cisplatin, 5-FU; - Cisplatin 75 (-100) mg/m²; - 5-FU 800 (-1000) mg/m²; Cisplatin / Capecitabine (XP); - Cisplatin 80 mg/m²; - Capecitabine 1000 mg/m²
  Arms: Arm B: Chemotherapy by Investigator's choice

SUMMARY:
The aim is to assess the relative efficacy of S-1 de-escalation therapy vs. continuation of chemotherapy after induction therapy in patients with metastatic esophagogastric cancer in terms of overall survival.

DETAILED DESCRIPTION:
Open-label, multi-center, controlled, randomized, parallel-group phase II trial in patients with metastatic esophagogastric cancer having received induction chemotherapy.

Patients will be registered before or after application of a three-months induction chemotherapy . This 12-week induction therapy will consist of one of the following regimens: FLO/mod. Folfox-6, Cisplatin/5-FU, Cisplatin/S-1, FLOT, EOX/EOF or XP. Regarding dose adjustments, Investigators should refer to Section 6.3 and to the summary of product characteristics of the chemotherapeutical agents. Patients having finished the preplanned induction therapy without tumor progression (i.e. with complete remission (CR), partial remission (PR), stable disease (SD) or non-CR/non-PD in patients with non-measurable disease only according to RECIST Criteria Version 1.1) at week 12, being able to swallow capsules and having Eastern Cooperative Oncology Group (ECOG) performance score of 0-1 will be randomized in a 2:1 ratio to receive Arm A or B.

In Arm A patients will continue with S-1 de-escalation phase starting at week 13 until disease progression, toxicities requiring discontinuation, withdrawal of consent, pregnancy, death or lost to follow up whichever occurs first. In patients with drug-related severe toxicity S-1 dose will be adjusted or study treatment will be terminated.

In Arm B patients will continue to receive the same polychemotherapy as during induction therapy until tumor progression, toxicities requiring discontinuation, withdrawal of consent, pregnancy, death or loss to follow up whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent incl. participation in translational research
2. Male or female patient 18 years or older
3. Histologically confirmed metastatic or locally advanced unresectable gastric adenocarcinoma or adenocarcinoma of the esophagus or the esophagogastric junction (Her-2/neu negative or with unknown Her-2/neu status)
4. Adjuvant/neoadjuvant or perioperative chemotherapy or (chemo-)radiotherapy must have been finished at least 6 months before start of the induction therapy
5. For patients enrolled before induction therapy: No previous systemic treatment (i.e. chemotherapy) for metastatic disease
6. For patients enrolled after induction therapy: Having finished a three-months induction therapy (6 cycles of a bi-weekly regimen, 4 cycles of a three-weekly regimens or 3 cycles of a four-weekly regimen) without tumor progression or limiting toxicity
7. ECOG Performance Score 0-1 (Karnofsky Performance status >= 80%)
8. Ability for oral intake of the study drug, patients with tumor-related problems with oral intake might be registered if the symptom is expected to be improved during induction therapy (e.g. due to a tumor stenosis)
9. Female patient of childbearing potential (i.e. did not undergo surgical sterilization - hysterectomy, bilateral tubal ligation, or bilateral oophorectomy - and is not post-menopausal for at least 24 consecutive months) with a negative pregnancy test
10. Hematology and biochemistry laboratory results within the limits normally expected for the patient population, defined by the following:

    * Absolute neutrophil count ≥ 1500/µl
    * Platelet count ≥ 100000/µl
    * Leukocyte count > 3000/µl
    * Hemoglobin ≥ 9 g/dL or 5.59 mmol/l, previous transfusions (>3 days) of erythrocytes are allowed
    * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), in patients with known Meulengracht syndrom ≤3 x ULN
    * AST ≤ 3xULN in absence of liver metastases, or ≤5xULN in presence of liver metastases
    * ALT ≤ 3xULN in absence of liver metastases, or ≤5xULN in presence of liver metastases
    * Creatinine clearance ≥30 mL/min according to Cockcroft-Gault formula

Exclusion Criteria:

1. Previous major sugery within the last 28 days before the start of the induction treatment. The implantation of a central venous access (e.g. porth-a cath system) is allowed.
2. History of other malignant tumors within the last 5 years before start of induction treatment, except basal cell carcinoma or curatively excised cervical carcinoma in situ
3. Known brain metastases
4. Concurrent radiotherapy involving target lesions used for this study. Concurrent palliative radiation for non-target lesions is allowed if other target lesions are available outside the involved field; previous radiotherapy including target lesions must have been finished at least 28 days before start of induction treatment.
5. For patients enrolled before the induction therapy: Previous systemic treatment (i.e. chemotherapy) for metastatic disease
6. Known active HBV, HCV infection or documented HIV infection
7. Serious concomitant disease or medical condition that by judgment of the Investigator renders the patient at high risk of treatment complications
8. Clinically relevant coronary artery disease (NYHA functional angina classification III/IV), congestive heart failure (NYHA III/IV), clinically relevant cardiomyopathy, history of myocardial infarction in the last 3 months, or high risk of uncontrolled arrhythmia
9. Female patient pregnant or breast feeding
10. Female patient of childbearing potential (i.e. did not undergo surgical sterilization - hysterectomy, bilateral tubal ligation, or bilateral oophorectomy - and is not post-menopausal for at least 24 consecutive months) not willing to use an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the end of treatment. Male patient not willing to use an adequate method of contraception to avoid conception throughout the study and for up to 26 weeks after the end of treatment in such a manner that the risk of pregnancy is minimized.
11. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 60 days prior to start of induction (e.g. one of the allowed standard chemotherapies (see above) with or without additional placebo within a clinical trial is allowed)
12. Chronic diarrhea or short bowel syndrome
13. Known hypersensitivity to S-1, other fluoropyrimidines or platinum compounds. Contraindication to receive S-1 or the polychemotherapy (induction & arm B) chosen for this patient as per current Summary of Product Characteristics. Known DPD deficiency
14. For patients enrolled before the induction therapy: Grade ≥2 peripheral neuropathy
15. Known drug abuse/alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2014-09; Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | approx. 12 month
  OS will be defined as the time length between randomization and the date of death from any cause or the date of last follow-up in case of no documentation of death.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | approx. 12 month
  PFS will be defined as the time length between the date of randomization and the date of first disease progression or death (whichever occurs first).
Quality of Life | approx. 12 month
  Quality of life will be evaluated using the validated European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 questionnaire and the gastric module STO22.

OTHER OUTCOMES:
Malnutrition | approx. 12 month
  Explorative descriptive statistical methods will be applied to describe the results of the Nutritional Risk Screening stratified by visit and treatment arm.
Overall Survival of non-randomized patients | approx. 12 month
  For exploratory purposes, the overall survival experience of non-randomized patients will be considered. The survival time is defined as the time length between start of induction therapy and the date of death from any cause or the date of last follow-up in case of no documentation of death.
Adverse Events | approx. 12 month
  For descriptive analysis of toxicity/safety, summary tables will be presented showing the total number of patients reporting at least one specific event stratified by System Organ Class, Common terminology criteria for adverse events (CTCAE) term, CTCAE grade and causality.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Martin Haag, Dr., Principal Investigator — NCT-Med. Onkologie
Locations (1):
- NCT-Med. Onkologie, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Stocker G, Lorenzen S, Ettrich T, Herz AL, Longo F, Kiani A, Venerito M, Trojan J, Mahlberg R, Moosmann N, Chibaudel B, Kubicka S, Greil R, Daum S, Geissler M, Larcher-Senn J, Keller G, Lordick F, Haag GM. S-1 maintenance therapy in Caucasian patients with metastatic esophagogastric adenocarcinoma-final results of the randomized AIO MATEO phase II trial. ESMO Open. 2023 Jun;8(3):101572. doi: 10.1016/j.esmoop.2023.101572. Epub 2023 Jun 2. PMID 37270871
- [Derived] Haag GM, Stocker G, Quidde J, Jaeger D, Lordick F. Randomized controlled trial of S-1 maintenance therapy in metastatic esophagogastric cancer - the multinational MATEO study. BMC Cancer. 2017 Jul 31;17(1):509. doi: 10.1186/s12885-017-3497-9. PMID 28760152
- See also: Working Group for Medical Oncology (AIO) from the German Cancer Society (DKG) — http://www.aio-portal.de